CLINICAL TRIAL: NCT04178356
Title: The Effects of Proprioceptive Neuromuscular Facilitation Training on Pain, Range of Motion, Functional Disability Index, Back Extensor Muscle Endurance, and Diaphragm Muscle Thickness in Patients With Chronic Low Back Pain
Brief Title: The Effects of Proprioceptive Neuromuscular Facilitation Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner Karartı, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019700
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Low Back Pain; Disability Physical
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Care Provider
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Study Group (Experimental): In addition to the conservative treatment of the control group, proprioceptive neuromuscular facilitation techniques will be applied for 4 weeks.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation Training
- Control Group (Active Comparator): Conservative treatment of low back pain will be applied for 4 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation Training — The Proprioceptive Neuromuscular Facilitation Training will be performed using patterns and techniques in various positions for abdominal and back muscles' facilitation and strengthening. Supine, side-lying, and sitting positions will be used. There will be a rest of about 20 sec between sets. Warm-up for 10 min, main exercises for 25 min, cool-down for 10 min (a total of 45 min), 5 times a week for 4 weeks.
  Arms: Experimental-Study Group
Other: Control Group — Ultrasound, TENS, massage, and exercise will be used with each other because in most of the physical therapy clinics these modalities are used together for such problems as a conventional treatment. After massage application, hamstring and paravertebral muscles stretching and also stabilizing exercises will be prescribed, each one for ten times in each session.
  Arms: Control Group

SUMMARY:
Although various methods have been emphasized in the treatment of chronic low back pain (CLBP), one of the treatments with the highest level of evidence is tailor-made exercises. Exercises to improve lumbopelvic region muscle performance and proprioception have been reported to be effective in alleviating clinical symptoms in individuals with CLBP. Proprioceptive neuromuscular facilitation (PNF) techniques are frequently used in the treatment of CLBP. PNF techniques reduce the load on vertebral bodies when performed in supine, side-lying, and sitting positions. It has been reported that performing a PNF trunk pattern in a sitting position is effective for treating CLBP and it improves muscle endurance, flexibility, and functional performance. PNF lower extremity pattern training in a supine position is effective for abdominal muscle activation. There is also an improvement in pain, functional disability, and fear-avoidance belief by applying the PNF coordination pattern in a standing position. While the diaphragm effect was emphasized in individuals with CLBP, no studies examining the effect of PNF techniques used on CLBP treatment on diaphragm muscle thickness were found. In addition, studies investigating the effect of PNF techniques on pain, functional disability index, range of motion and waist muscle endurance were found to be insufficient. Therefore, the aim of this study was to investigate the effect of PNF techniques on related variables in individuals with CLBP.

DETAILED DESCRIPTION:
It is known that dorsal proprioceptive signals, one of the necessary components in providing lumbopelvic motor control, are decreased in individuals with chronic low back pain (CLBP) and respiratory dysfunction. Diaphragm, which is an important postural control muscle, plays an important role in the correct reception of these signals. Electromyographic and ultrasonographic measurements in healthy subjects showed that the diaphragm was activated for anticipatory automatic adjustments before shoulder flexion, adjusted the transdiaphragmatic pressure and shortened the neck before motion began. In CLBP, diaphragm motility decreases significantly due to fatigue in the diaphragm. This makes it difficult to perform anticipatory automatic arrangements, leading to postural instability and respiratory dysfunction. Although various methods have been emphasized in the treatment of CLBP, one of the treatments with the highest level of evidence is tailor-made exercises. Exercises to improve lumbopelvic region muscle performance and proprioception have been reported to be effective in alleviating clinical symptoms in individuals with CLBP. Proprioceptive neuromuscular facilitation (PNF) techniques are frequently used in the treatment of CLBP. PNF techniques reduce the load on vertebral bodies when performed in supine, side-lying, and sitting positions. It has been reported that performing a PNF trunk pattern in a sitting position is effective for treating CLBP and it improves muscle endurance, flexibility, and functional performance. PNF lower extremity pattern training in a supine position is effective for abdominal muscle activation. There is also an improvement in pain, functional disability, and fear-avoidance belief by applying the PNF coordination pattern in a standing position. While the diaphragm effect was emphasized in individuals with CLBP, no studies examining the effect of PNF techniques used on CLBP treatment on diaphragm muscle thickness were found. In addition, studies investigating the effect of PNF techniques on pain, functional disability index, range of motion and waist muscle endurance were found to be insufficient. Therefore, the aim of this study was to investigate the effect of PNF techniques on related variables in individuals with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* presence of non-spesific CLBP (˃3 months),
* the ability to understand and follow verbal commands,
* to be volunteer to participate in the study.

Exclusion Criteria:

* to be pregnant,
* had a previous history of spinal surgery,
* neurological deficits,
* specific LBP (including facet joint syndrome, disc herniation and sacroiliac joint dysfunction),
* cancer or other autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 4 weeks
  The pain severity of the patients with CLBP will be measured using a 10 centimeter VAS where score of 0/10 indicated no pain and 10/10 to indicated intolerable pain, respectively. A clinically meaningful difference for the VAS is a reduction of approximately two points for patients with CLBP.

SECONDARY OUTCOMES:
The Oswestry Disability Index (ODI) | 4 weeks
  This scale is intended to measure the disability level due to CLBP. It consists of ten questions: pain intensity, personal care, lifting, walking, sitting, standing, sleep¬ing, sex life, and social life. Depending on performance ability, 6 levels (0 to 5 points) can be specified: the higher the score, the greater the disability. The ODI is calculated by dividing the total score by the number of questions answered and multiplying by 100. The participants will be asked whether any statements characterized them on evaluation day. The Turkish version of ODI has good comprehensibility, internal consistency, and validity and is an adequate and useful instrument for the assessment of disability in patients with low back pain (internal consistency=0.89-0.91). The minimal detectable change on the ODI is 6-10 points. Clinically meaningful change is considered to be 30-50%.
The Schober Test | 4 weeks
  The Schober Test will be used for the assessment of lumbar flexion range of motion (ROM) of the patients with CLBP. In relaxed standing position, the mid-point between the two posterior superior iliac spines will be determined. Then, 5 centimeter above and 5 centimeter below this point will be marked as measurement points. At this stage, patients will be asked to bend forwardly as much as possible while maintaining their knees as straight as possible. The difference between the two points in this position in comparison to distance between the points in relaxed standing position will be considered as the lumbar flexion ROM.
The Prone Doubled Leg Straight Leg Raising (SLR) | 4 weeks
  SLR will be used for the evaluation of back extensor muscle endurance of the patients with CLBP. Participants lay in prone position with their hips extended, putting their hands underneath their foreheads. They will be asked to raise both of their legs until knee clearance will be achieved. At this stage the examiner will record the time until the participant will no longer able to keep knee clearance. The recorded time in seconds will be considered as back extensor muscle endurance.
Ultrasonographic Imaging | 4 weeks
  Ultrasonographic imaging will be conducted by a radiologist (experience˃15 years) to determine muscle thickness of diaphragm. Thickness of both hemidiaphragm will be measured at the end of expiration from transvers and sagittal images obtained at the 9th intercostal space on anterior axillary line.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Beeckmans N, Vermeersch A, Lysens R, Van Wambeke P, Goossens N, Thys T, Brumagne S, Janssens L. The presence of respiratory disorders in individuals with low back pain: A systematic review. Man Ther. 2016 Dec;26:77-86. doi: 10.1016/j.math.2016.07.011. Epub 2016 Jul 25. PMID 27501326
- [Result] Areeudomwong P, Wongrat W, Neammesri N, Thongsakul T. A randomized controlled trial on the long-term effects of proprioceptive neuromuscular facilitation training, on pain-related outcomes and back muscle activity, in patients with chronic low back pain. Musculoskeletal Care. 2017 Sep;15(3):218-229. doi: 10.1002/msc.1165. Epub 2016 Oct 28. PMID 27791345
- [Result] Kofotolis N, Kellis E. Effects of two 4-week proprioceptive neuromuscular facilitation programs on muscle endurance, flexibility, and functional performance in women with chronic low back pain. Phys Ther. 2006 Jul;86(7):1001-12. PMID 16813479